CLINICAL TRIAL: NCT05605132
Title: Comparison of the Effects of Proprioception and Tactile Accuracy Training on Proprioception, Range of Motion, Pain and Disability in Patients With Chronic Neck Pain
Brief Title: SENSORY RE-TRAINING IN PATIENTS WITH CHRONIC NECK PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Canli, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neck Pain
Record Dates: First submitted 2022-10-29; First posted 2022-11-04 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2022-11

CONDITIONS: Neck Pain; Cervical Pain; Neck Muscle Issue; Neck Pain, Posterior; Cervical Pain, Posterior
Keywords: oculomotor exercises; neck pain; cervical pain; sensory re-training
MeSH Terms: conditions — Neck Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioceptive Training Group (Experimental): oculomotor exercises will be applied to the participants three times a week for four weeks.
  oculomotor exercises:
  head relocation gaze stability eye follow saccadic eye movement head and eye coordination
  Interventions: Other: Proprioceptive Training Exercise
- Tactile Acuity Training (Experimental): Participants will be requested to lie face down. Five points will be marked in the painful areas on the right and left sides of the neck. The distance between the points will equal the two-point discrimination value. A photograph of the neck will be taken. The patient will not see his/her own neck during the application but see the photograph of his/her neck. The points will be touched lightly with two different stimuli (a pen with a 2 mm diameter and a mushroom probe with an 11 mm diameter). Participants will be asked about the location and type of the stimuli. The interstimulus interval will be 15 seconds. If more than 90% of correct answers are obtained, the distance between the points will be reduced by 10%. The training will be performed in three separate blocks, a total of 72 stimuli (block duration = 6 minutes, rest time between blocks = 3 minutes, number of stimuli applied in each block = 24 stimuli). The treatment time will be 24 minutes.
  Interventions: Other: Tactile Acuity Training
- Control Group (Sham Comparator): The participants will be evaluated two times at 4-week intervals. No intervention will be applied during the time frame.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Proprioceptive Training Exercise — oculomotor exercises will be applied to the participants three times a week for four weeks.
  oculomotor exercises:
  * head relocation
  * gaze stability
  * eye follow
  * saccadic eye movement
  * head and eye coordination
  Arms: Proprioceptive Training Group
Other: Tactile Acuity Training — Participants will be requested to lie face down. Five points will be marked in the painful areas on the right and left sides of the neck. The distance between the points will equal the two-point discrimination value. A photograph of the neck will be taken. The patient will not see his/her own neck during the application but see the photograph of his/her neck. The points will be touched lightly with two different stimuli (a pen with a 2 mm diameter and a mushroom probe with an 11 mm diameter). Participants will be asked about the location and type of the stimuli. The interstimulus interval will be 15 seconds. If more than 90% of correct answers are obtained, the distance between the points will be reduced by 10%. The training will be performed in three separate blocks, a total of 72 stimuli (block duration = 6 minutes, rest time between blocks = 3 minutes, number of stimuli applied in each block = 24 stimuli). The treatment time will be 24 minutes.
  Arms: Tactile Acuity Training
Other: Control Group — The participants will be evaluated two times at 4-week intervals. No intervention will be applied during the time frame.
  Arms: Control Group

SUMMARY:
It is known that tactile acuity and proprioceptive sense decrease in patients with chronic neck pain. However, sensory re-training in patients with chronic neck pain has not been given sufficient importance. The effects of proprioceptive and tactile acuity training on pain intensity in patients with chronic neck pain will be compared in this study. Eligible participants will be divided into three groups as follows: Proprioceptive Training Group (PTG), Tactile Acuity Training Group (TAG), and Control Group (CG). The randomization will be performed using the block randomization method to obtain an equal number of participants in the groups. Each participant will be evaluated two times at a 4-week interval. Participants will be evaluated regarding subjective pain intensity by using a Numerical Rating Scale, temporal summation, and conditioned pain modulation using an algometer (JTECH Medical-Algometer Commander, USA). Neck proprioception exercises will be applied to the patients in the PTG at 3 days a week for 4 weeks. Tactile acuity training will be applied to the patients in the TAG 3 days a week for 4 weeks. Between the two assessments, the Control Group will not receive any treatment.

ELIGIBILITY:
Inclusion Criteria:

* to be aged between 20-60 years old
* Pain limited to the posterior of the cervical region.
* Pain that lasts longer than 3 months
* Pain severity of 3 or higher on the Visual Analog Scale

Exclusion Criteria:

* Malignant tumor in any part of the body (no screening will be performed for the presence of tumor and patients diagnosed with tumors before the study will not be included).
* Vertebral fractures
* Fibromyalgia
* chronic fatigue syndrome
* History of surgery in the neck or shoulder area
* Radicular pain
* Neurological deficit of disc pathologies
* Spinal stenosis
* Spondylolisthesis
* Pronounced cervical kyphosis
* Significant scoliosis involving the cervical region

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | Change form baseline at 4 weeks
  It will be evaluated using a Numerical Rating Scale (0 indicate no pain, 10 indicate most vulnerable pain)

SECONDARY OUTCOMES:
pressure pain threshold | Change form baseline at 4 weeks
  It will be evaluated in the middle of the upper trapezius muscle and the dominant side of the tibialis anterior muscle. It will be evaluated two times at 30-second intervals. The average of value will be recorded.
temporal summation | Change form baseline at 4 weeks
  It will be evaluated in the middle of the upper trapezius muscle. 10 subsequent stimuli with a 1-second application at the level of pressure pain threshold and 1-second rest. Pain intensity at 1, 5 and 10th stimuli will be asked based on the Numerical Rating Scale.
conditioned pain modulation | Change form baseline at 4 weeks
  The sphygmomanometer will be applied on the arm which is the contralateral side of the upper trapezius. It will be inflated at a rate of 20 mm/Hg and held at this value for 30 seconds. Then, the patient's pain intensity will be questioned according to the numerical pain scale.
neck disability | Change form baseline at 4 weeks
  A neck disability questionnaire (NDI) will be used

CONTACTS AND LOCATIONS:
Overall Officials: Kübra canlı, Study Chair — Hacettepe University; Filiz Can, Study Director — Hacettepe University; Gökhan Demirkıran, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe Universty, Ankara, Sıhhıye
  - Kübra, Ankara, Sıhhıye

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canli K, Demirkiran G, Can F. The efficiency of tactile discrimination training and oculomotor exercises in people with chronic neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2025 May 27;26(1):519. doi: 10.1186/s12891-025-08755-0. PMID 40420069